CLINICAL TRIAL: NCT01043978
Title: Prevention of Overfeeding During Infancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 200715679
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Novel nipple (Experimental)
  Interventions: Behavioral: Use of baby bottle nipple
- Coventional nipple (Active Comparator)
  Interventions: Behavioral: Use of baby bottle nipple

INTERVENTIONS:
Behavioral: Use of baby bottle nipple — Participants will be assigned to either a novel nipple or a conventional nipple to use when feeding their infants with the bottle

SUMMARY:
The overall goal of this project is to identify strategies to prevent overfeeding during infancy. One objective is to evaluate the impact on intake of allowing the infant greater control over the amount consumed when feeding from a bottle. This will be accomplished via the use of a novel nipple that mimics (functionally) the nipple of a human breast and allows the infant to self-regulate milk flow. The second objective is to evaluate the relationship between parental feeding styles and infant intake.

ELIGIBILITY:
Inclusion Criteria:

* Infant born at > 37 weeks gestation
* Infant weighed >2500 g at birth
* Infant is apparently healthy
* Mother speaks English
* Mother is 18 years of age or older
* Mother/infant pair lives within a 10-mile radius around the UC Davis Medical Center in Sacramento, CA
* Mother plans to use a bottle (at least occasionally) to feed her infant before he/she is 3 months old.

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 231 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Intake | per feed

SECONDARY OUTCOMES:
Growth | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn G Dewey, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States